CLINICAL TRIAL: NCT02198196
Title: Mind/Body Stress Management to Improve Outcomes in Workplace Weight Loss Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AT007845-01A1 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight Talk-Mindfulness (Experimental): WT-M retain the evidence-based elements of WT-S (control condition), including the DASH diet, physical activity components, and an emphasis on self-monitoring. However, each call in WT-M will include an emphasis on mindfulness and stress management that will not be included in the control condition.
  Interventions: Behavioral: Weight Talk-Mindfulness
- Weight Talk-Standard (No Intervention): Weight Talk-Standard is a phone and web-based weight loss intervention offered by employers as a benefit to their employees. Weight Talk is based on the NIH Clinical Guidelines on Identification, Evaluation and Treatment of Overweight and Obesity in Adults and utilizes the curriculum developed for the Diabetes Prevention Program. Weight Talk-S contains no additional stress management techniques.

INTERVENTIONS:
Behavioral: Weight Talk-Mindfulness
  Arms: Weight Talk-Mindfulness

SUMMARY:
The purpose of this study is to explore the efficacy of a phone-based weight loss program that has stress management techniques integrated throughout (Weight Talk-Mindfulness). The program is targeted at employees of certain companies who meet a cut-off score on a measure of stress-related eating. The control group will receive a standard phone-based program with no additional stress management information (Weight Talk-Standard).

* Hypothesis 1: Participants in Weight Talk-Mindfulness (WT-M; n=50) will experience decreases in their stress-related & emotion-related eating compared to the Weight Talk-Standard (WT-S; n=25) group.
* Hypothesis 2: The WT-M group will lose more weight compared to the WT-S control group.
* Hypothesis 3: Participants in WT-M will experience decreased perceived stress, increased eating self-efficacy, increased acceptance of weight-related thoughts & feelings and increased mindfulness compared to those in the WT-S control arm.
* Hypothesis 4: Participants in WT-M will be equally as satisfied with their weight loss program as those in WT-S.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in the Weight Talk program, inclusion criteria:

  * Employment by one of the employers who contract for Weight Talk services
  * Being over 18 years of age
  * Speak and read English
* Have a starting BMI between 25 and 35.
* Score 5 or higher on the 8-item Internal Disinhibition subscale of the Eating Inventory.
* Have regular access to email and internet.
* Willingness and ability to complete study and intervention procedures, including completing assessments, engaging in moderate physical activity (e.g., walking, swimming) and using the electronic scale at least once per week.

Exclusion Criteria:

* Type 2 Diabetes (Type 1 is an exclusion for the Weight Talk program).
* Past diagnosis of anorexia nervosa or bulimia nervosa.
* Weight Talk program exclusion criteria include:

  * Pregnancy
  * Bariatric surgery within past 12 months or planned in the next 6 months
  * Undergoing dialysis
  * Have Type 1 Diabetes diagnosis
* Women who are pregnant are not eligible for the program, but contraception is not required as this is a low risk study
* Currently using or planning to start using a pharmaceutical weight loss drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Eating Inventory - Internal Disinhibition subscale | Screening and 6-month follow-up
  8 items, screens for emotion and stress-related eating habits

SECONDARY OUTCOMES:
Body weight | Screening and 6-month follow-up
  Weight in pounds

OTHER OUTCOMES:
Mindful Eating Questionnaire | Screening, 6-month follow-up
  28-item scale that measures non-judgmental awareness of physical and emotional sensations associated with eating.
Rapid Fruit and Vegetable Screener | Screening, 6-month follow-up
  10-item scale that assesses fruit and vegetable intake.
Fat Screener | Screening, 6-month follow-up
  17-item scale that assesses fat intake
Sweets Eating | Screening, 6-month follow-up
  2-item scale that assesses high sugar food and drink intake
Perceived Stress Scale - 4 item | Screening, 6-month follow-up
  a 4-item scale that evaluates the appraisal of stress in one's life
Binge Eating Scale | Screening, 6-month follow-up
  16-item scale that assesses the presence of binge eating behaviors.
Behavioral Obesity Phenotype Scale | Screening, 6-month follow-up
  8-item scale that assesses lack of control, lack of satiation, and preoccupation with food. We include 6 out of the 8 original items; 2 of the items already exist in the Binge Eating Scale (BES). One additional Preoccupation with Food item was added.
Acceptance and Action Questionnaire for Weight Related Difficulties | Screening, 6-month follow-up
  22-item scale that measures acceptance and flexibility in relation to problematic thoughts and feelings regarding weight.
Generalized Anxiety Disorder scale | Screening, 6-month follow-up
  7-item diagnostic scale that assesses an individual's severity of anxiety and is used as a clinical screening tool for generalized anxiety disorder.
Personal Health Questionnaire | Screening, 6-month follow-up
  2-item scale that assesses the frequency of depressed mood over the past 2 weeks and is used as a preliminary screening tool for depression.
Adapted Physical Activity Measure | Screening, 6-month follow-up
  11-item scale that assesses overall activity level over the past week, adapted from measure used in the National Health and Nutrition Examination Survey (NHANES)
Five Facet Mindfulness Questionnaire: Short Form | Screening, 6-month follow-up
  24-item scale that measures non-judgmental awareness of thoughts, feelings, and physical sensations.
Satisfaction and Adherence | 6-month follow-up
  11-item measure consisting of Likert scale and open-ended questions about the participants' experience with the intervention and their adherence to mindfulness practice assignments.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Alekel, PhD, Study Chair — National Center for Complementary and Integrative Health (NCCIH); Kelly Carpenter, PhD, Principal Investigator — Consumer Wellness Solutions; Jennifer Lovejoy, PhD, Principal Investigator
Locations (1):
- Alere Wellbeing, Inc, Seattle, Washington, United States